CLINICAL TRIAL: NCT03076255
Title: A Single Institution Pilot Study Using a Head and Neck Maskless Immobilization Device (MID) for Patients With Head and Neck Cancer or Intracranial Tumors
Brief Title: Using a Head and Neck Maskless Immobilization Device For Patients With Intracranial Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16D.557; JT 8994 (Other: JeffTrial Number)
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Brain and Nervous System; Intracranial Neoplasm; Head and Neck Cancer
MeSH Terms: conditions — Neurologic Manifestations; Brain Neoplasms; Head and Neck Neoplasms | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Supportive care (MID) (Experimental): Patients undergo Computed Tomography (CT) simulation with thermoplastic mask and maskless immobilization device (MID) for radiation therapy (RT) planning on day 1. Patients undergo standard of care RT using thermoplastic mask only and cone-beam computed tomography (CBCT) imaging with thermoplastic mask and MID on day 8 and 15.
  Interventions: Procedure: Computed Tomography; Device: Medical Device; Procedure: Cone-Beam Computed Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT simulation
  Other Names: CAT Scan; CAT; Computerized Axial Tomography
Device: Medical Device — Given thermoplastic mask
Device: Medical Device — Given MID
Procedure: Cone-Beam Computed Tomography — Undergo CBCT imaging

SUMMARY:
This pilot clinical trial studies how well head and neck maskless immobilization device works in immobilizing patients with head and neck cancers or intracranial tumors undergoing radiation therapy. Maskless immobilization device may help to prevent movement of head during radiation therapy and immobilize patients with the same accuracy and reliability as the standard thermoplastic mask routinely used for patients receiving radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the setup accuracy and reproducibility of the maskless immobilization device (MID) in patients being treated for head and neck cancers or intracranial tumors who require radiation therapy

SECONDARY OBJECTIVES:

I. To assess the patient comfort and quality of life with the MID compared to the thermoplastic mask.

ELIGIBILITY:
Inclusion Criteria:

* Patients being treated for head and neck cancers who require radiation therapy or intracranial tumors, over a 2 to 7 week period of time
* Age ≥ 18 years old
* Subjects are capable of giving informed consent or have an acceptable surrogate capable of giving consent on the subject's behalf
* Provide signed and dated informed consent form

Exclusion Criteria

* History of prior trauma or orthopedic surgery to the cervical vertebral column/spine, which may interfere with the RT planning process
* Patient requires a neck brace for medical reasons
* Skull or bony defect in the area contacting the immobilization straps
* RT delivered by clinical setup only (no CT simulation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Voichita Bar Ad, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive care (MID)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Supportive care (MID)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11
  Hispanic or Latino | 1

OUTCOME MEASURES:

1. Primary Outcome: Accuracy Measured by Quantifying the Difference in Translational Shifts From the Daily Setup to Planning CT Scan Digitally Reconstructed Radiograph
Description: The primary endpoints are to assess the setup accuracy and reproducibility with the Maskless Immobilization Device. Accuracy will be measured by quantifying the difference in translational shifts from the daily setup to planning CT scan digitally reconstructed radiograph (DRR). The magnitude of shifts will be compared to the shifts required using the gold standard thermoplastic mask. Translational shifts is defined as measuring the shifts in cm between the daily setup and the planning setup.
Time Frame: Baseline to Day 15, an average of 31 days
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Supportive care (MID)
Number analyzed (Participants) | 12
centimeters (cm)
  Vertical | 0.08 (0.30)
  Longitudinal | 0.16 (0.52)
  Lateral | -0.02 (0.47)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from day 1 of participation, at visit 2 (day 8 +/- 5 days), at visit 3 (day 15 +/- 5 days) and at 7 days after the last day of study participation.
Description: An adverse event is any untoward or unfavorable medical occurrence in a human subject, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the subject's participation in the research, whether or not considered related to the subject's participation in the research.
Arm/Group | Supportive care (MID)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive care (MID) (N=12)
Hyperglycemia - Grade IV (Endocrine disorders) | 1 (1)
DKA (Endocrine disorders) | 1 (1)
Dehydration - Grade 3 (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive care (MID) (N=12)
depression (Psychiatric disorders) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1)
obstructive sleep apnea (Reproductive system and breast disorders) | 1 (1)
headache (General disorders) | 3 (3)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Lymphedema (Blood and lymphatic system disorders) | 1 (1)
hypertension (Vascular disorders) | 4 (4)
Tachycardia (Cardiac disorders) | 2 (2)
Visual Disturbance (Eye disorders) | 2 (2)
Optic Nerve Disorder (Eye disorders) | 1 (1)
Tremor (Nervous system disorders) | 4 (4)
Seizure (Nervous system disorders) | 3 (3)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Cerebral Edema (Nervous system disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Ulnar neuropraxia (Nervous system disorders) | 1 (1)
watering eyes (Eye disorders) | 1 (1)
Flat Affect (Psychiatric disorders) | 1 (1)
Erythema (abdomen) (Skin and subcutaneous tissue disorders) | 1 (1)
Scar Weeping (Skin and subcutaneous tissue disorders) | 1 (1)
Right upper extremity weakness (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Weight loss (Metabolism and nutrition disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Papular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1)
Floppy eyelid syndrome (Eye disorders) | 1 (1)
Chronic venous stasis (Vascular disorders) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 4 (4)
Abnormal Urine Culture (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Hypocalcemia (Renal and urinary disorders) | 1 (1)
Hypermagnesemia (Renal and urinary disorders) | 1 (1)
INR increased (Blood and lymphatic system disorders) | 1 (1)
increased appetite (Metabolism and nutrition disorders) | 1 (1)
fatigue (General disorders) | 6 (6)
apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood in stool (Gastrointestinal disorders) | 1 (1)
rectal pain (Gastrointestinal disorders) | 1 (1)
ALP increased (Hepatobiliary disorders) | 1 (1)
Paresthesia (Skin and subcutaneous tissue disorders) | 2 (2)
Diaphoretic (Skin and subcutaneous tissue disorders) | 1 (1)
hemorrhagic per-rectal abscess (Infections and infestations) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysosmia (General disorders) | 1 (1)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 4 (4)
Alopecia (Immune system disorders) | 3 (3)
Hypernatremia (Blood and lymphatic system disorders) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
lymphocyte count decreased (Blood and lymphatic system disorders) | 2 (2)
esophageal pain (General disorders) | 1 (1)
Insomnia (General disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Bruises easily (Blood and lymphatic system disorders) | 1 (1)
Dysarthria (General disorders) | 3 (3)
Paresthesia (Nervous system disorders) | 1 (1)
Skin color change (Skin and subcutaneous tissue disorders) | 1 (1)
Hearing impairment (Ear and labyrinth disorders) | 1 (1)
Hand cramping (Musculoskeletal and connective tissue disorders) | 2 (2)
Cognitive disturbance (Psychiatric disorders) | 1 (1)
Nevi (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Cracked tooth (Injury, poisoning and procedural complications) | 1 (1)
Diabetes Mellitus (Endocrine disorders) | 2 (2)
Left hand disability (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperlipidemia (Blood and lymphatic system disorders) | 1 (1)
Ataxia (General disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Delirium (Congenital, familial and genetic disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Pain - incision site (Surgical and medical procedures) | 2 (2)
nausea/vomiting (General disorders) | 1 (1)
hypocholesteremia (Blood and lymphatic system disorders) | 1 (1)
Ear pain (General disorders) | 1 (1)
Apathy (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT03076255/Prot_SAP_000.pdf